CLINICAL TRIAL: NCT04358796
Title: Measuring Cognitive Enhancement During Hyperbaric Oxygen Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Shay Efrati, Medical Director of the Sagol Center for Hyperbaric Medicine, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0031-17-ASF
Record Dates: First submitted 2020-02-09; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Hyperbaric Oxygen Therapy
Keywords: Cognitive enhancement; Memory; Information processing speed; Hyperbaric oxygen treatments

STUDY DESIGN:
Intervention Model Description: two groups being tested in parallel. The first group in HBOT environment. The second group in a SHAM environment.
Who Masked: Participant
Masking Description: Patients are unaware to the ATA in chamber and to oxygen levels in their mask.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HBOT environment (Experimental): Cognitive testing in 2ATA, 100% oxygen in breathing-masks
  Interventions: Device: Hyperbaric oxygent treatment
- Control environment (Sham Comparator): Cognitive testing in 1ATA, air in breathing-masks
  Interventions: Device: Control hyperbaric oxygen treatment

INTERVENTIONS:
Device: Hyperbaric oxygent treatment — Subjects will enter the oxygen chamber. ATA will be elevated to 2 ATA. They will breath 100% oxygen while solving cognitive tests designed to assess their cognitive capacities
  Arms: HBOT environment
Device: Control hyperbaric oxygen treatment — Subjects will enter the oxygen chamber. ATA will be elevated to 1.2 ATA for a short while and the decreased back to 1 ATA. They will breath air while solving cognitive tests designed to assess their cognitive capacities
  Arms: Control environment

SUMMARY:
The aim of the current study was to examine the effect of short-term HBOT (hyperbaric oxygen treatments) on a range of cognitive abilities. The current study examined whether there is a HBOT-related short-term cognitive improvement and, if so, what specific cognitive abilities are improved by the intervention.

Participants were randomized to perform cognitive tasks in one of two chambers with two different clinical environments: (a) HBOT condition: (2 ATA (atmosphere absolute) 100% oxygen for 90 minutes). (b) Control condition: in which the chamber was not pressurized (Normobaric condition- 1 ATA for 90 minutes).

DETAILED DESCRIPTION:
The aim of the current study was to examine the effect of short-term HBOT on a range of cognitive abilities. The current study examined whether there is a HBOT-related short-term cognitive improvement and, if so, what specific cognitive abilities are improved by the intervention.

Participants were recruited through ads on the internet and on student social groups. All participants underwent a comprehensive physical and neurological examination, and general medical conditions were ruled out. Participants were excluded if reported changes in their cognitive or behavioral functions during one month prior to the beginning of the study. Smokers (people who smoke more than seven cigarettes a week) were required to take a lung x-ray confirming there isn't a pulmonary pathology, such as pneumothorax, pulmonary bullae, emphysema, or other lung pathologies preventing them from staying in a high ATA environment. Participants with an abnormal x-ray were excluded from the study. Participants who regularly use Methylphenidate (i.e. Ritalin) or other stimulants for attention disorders (i.e. ADHD) were instructed not to take it at the day of the experiment.

Following consent, all the participants were exposed to the testing battery in a group setting. One of the experimenters went through each of the sub-tests instructions in a detailed manner prior to a practice phase in which participants trained on the tasks. Afterwards, participants were randomized to perform the tasks in one of two chambers with two different clinical environments: (a) HBOT condition: (2 ATA 100% oxygen for 90 minutes). The atmospheric pressure in this condition was set to 2 ATA. This ATA level is known to have a clinical effect, whereas higher-pressure levels may result in inhibitory brain effects or even lead to focal toxicity (Efrati and Ben-Jacob, 2014). (b) Control condition: in which the chamber was not pressurized (Normobaric condition- 1 ATA for 90 minutes) and participants breathed air (21% oxygen). In this condition, ATA was elevated for a few minutes to 1.2 ATA in order to mimic the feeling of pressure building up in the ears. The pressure was decreased soon after to 1 ATA.

The assessment began 30 min after participants wore the oxygen masks within the chamber, in order to enable appropriate brain oxygenation in the HBOT condition (Vadas et al., 2017). The battery was composed of cognitive tests adapted for high functioning subjects and adjusted to an in-chamber group administration setting.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-40
* intact sight / corrected sight
* Hebrew as mother tongue
* Intact comprehension

Exclusion Criteria:

* Active neurologic or psychiatric diagnosis.
* If Had been treated with HBOT for any other reason prior to their inclusion;
* Chest pathology ;
* Inner ear disease;
* Claustrophobia;

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
memory | after 20 minutes of intervention
  Number of words retrieved from a list
Working memory | after 20 minutes of intervention
  accuracy rates on a working memory paradigm (n-back)
Divided attention | after 20 minutes of intervention
  accuracy rates on a divided attention task (identifying visual and auditory targets)
Information processing speed | after 20 minutes of intervention
  Accuracy rates on an information processing speed task (Symbol tracing task)
Response inhibition | after 20 minutes of intervention
  Accuracy rates on a response inhibition task (stroop)
Problem solving | after 20 minutes of intervention
  accuracy rates on a problem solving task (solving arithmetic series)

CONTACTS AND LOCATIONS:
Overall Officials: Shay Efrati, Study Director — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No